CLINICAL TRIAL: NCT05366816
Title: ctDNA-Guided Sunitinib And Regorafenib Therapy for Gastrointestinal Stromal Tumor (GIST)
Brief Title: ctDNA-Guided Sunitinib And Regorafenib Therapy for GIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jonathan Trent, MD, PhD, Professor of Clinical, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20201368
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: KIT Exon 13 receiving Sunitinib (Experimental): Participants with KIT mutation on exon 13 will receive Sunitinib. Participants showing disease progression after first-assigned Sunitinib therapy have the option to receive Regorafenib therapy. Total allotted time for treatment is up to 12 months.
  Interventions: Drug: Sunitinib; Drug: Regorafenib
- Group B: KIT Exon 17 receiving Regorafenib (Experimental): Participants with KIT mutation on exon 17 will receive Regorafenib. Participants showing disease progression after first-assigned Regorafenib therapy have the option to receive Sunitinib therapy. Total allotted time for treatment is up to 12 months.
  Interventions: Drug: Sunitinib; Drug: Regorafenib

INTERVENTIONS:
Drug: Sunitinib — 37.5 mg of Sunitinib orally (PO), once daily on a 28-day treatment cycle.
  Other Names: Sutent; SU11248
Drug: Regorafenib — 120.0 mg of Regorafenib, once daily by mouth 3 weeks on 1 week off on a 4-week treatment cycle.
  Other Names: Stivarga; Regonix; BAY 73-4506

SUMMARY:
The purpose of this research is to test if mutations (changes in DNA) in exons (segment of DNA or RNA containing information that has the instructions for making proteins) in the KIT gene can be used to predict the body's response to standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥ 18 years of age.
2. Patients who have histologically confirmed metastatic or unresectable GIST. Unresectable GIST must be confirmed to be unresectable by an experienced surgeon.
3. Patients who received imatinib prior treatment regimens, including adjuvant therapy, with objective disease progression, inadequate clinical benefit, or intolerance. Additionally, disease progression or intolerance to other systemic therapies including investigational agents and radiotherapy is allowed. Patients who experienced intolerance to prior therapies must have objective disease progression prior to enrollment.
4. Patients who have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2.
5. Patient, or legal guardian if permitted by local regulatory authorities, who provides informed consent to participate in the study.
6. Presence of proto-oncogene c-KIT (KIT) exon 13 or 17 secondary mutation will be determined through a circulating tumor DNA (ctDNA) blood test or biopsy performed as per standard of care.

Exclusion Criteria:

1. Patients who have received prior treatment with sunitinib or regorafenib.
2. Patients who have received more than 2 different prior tyrosine kinase inhibitor (TKI) treatment regimens. If a patient receives the same TKI more than once sequentially (eg, imatinib followed by a period without systemic therapy and retreatment with imatinib), that will be counted as a single TKI treatment regimen.
3. Patients who are known to be KIT wild type.
4. Patients who received any systemic anticancer therapy within 2 weeks before. Prior radiotherapy to major organs within 2 weeks of admission, or focal radiotherapy, such as to bones, limbs, or other areas not involving major organs, within 3 days.
5. Patients who have clinically significant, uncontrolled, cardiovascular disease, including congestive heart failure Grades II, III or IV according to the New York Heart Association classification, myocardial infarction or unstable angina within the previous 6 months, or uncontrolled hypertension.
6. Patients who have experienced arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within the 6 months before randomization or venous thrombotic events such as deep vein thrombosis within the 3 months before screening.
7. Patients who have experienced any hemorrhage or bleeding event NCI CTCAE version 5.0 Grade 3 or higher within 4 weeks before screening.
8. Patients who have a known risk of intracranial bleeding, such as a brain aneurysm or history of intracranial bleeding within 1 year prior to screening.
9. Patients who have a non-healing wound, ulcer, or bone fracture.
10. Patients who have poor organ function as defined by one or more of the following laboratory parameters:

    * Persistent proteinuria of NCI-CTCAE version 4.03 Grade 3 or higher
    * Alanine aminotransferase and aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN) if no hepatic metastases are present; > 5 × ULN if hepatic metastases are present.
    * Total bilirubin >1.5 × ULN; and in presence of Gilbert's syndrome, total bilirubin > 3 × ULN or direct bilirubin > 1.5 × ULN.
    * Estimated (Cockcroft-Gault formula) or measured creatinine clearance < 40 mL/min.
    * Platelet count < 90 × 109/L and absolute neutrophil count (ANC) < 1.0 × 10^9/L.
    * Hemoglobin < 9 g/dL. Transfusion and erythropoietin may be used to reach at least 9 g/dL, but must have been administered at least 2 weeks before screening.
11. Patients who have received neutrophil growth factor support within 14 days of screening.
12. Patients who require therapy with a concomitant medication that is a strong inhibitor or strong inducer of CYP3A4.
13. Patients who have had a major surgical procedure (minor surgical procedures such as central venous catheter placement, tumor needle biopsy, and feeding tube placement are not considered major surgical procedures) within 14 days of screening. Patient has significant traumatic injury within 28 days before screening.
14. Patients who have a history of another primary malignancy that has been diagnosed or required therapy within 2 years before screening. (The following are exempt from the 2-year limit: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate cancer, and completely resected carcinoma in situ of any site.)
15. Patients who have a history of a seizure disorder requiring anti-seizure medication.
16. Patients who have metastases to the brain.
17. Patients who are unwilling or unable to comply with scheduled visits, drug administration plan, laboratory tests, or other study procedures and study restrictions.
18. Patients who have a QT interval corrected using Fridericia's formula (QTcF) of > 450 msec.
19. Women who are unwilling, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of randomization and for at least 30 days after the last dose of study drug. Men who are unwilling, if not surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of randomization and for at least 90 days after the last dose of study drug. Refer to Appendix G for acceptable methods of contraception.
20. Women who are pregnant, as documented by a serum beta human chorionic gonadotropin (β-hCG) pregnancy test consistent with pregnancy, obtained within 7 days before the treatment assignment. Females with β-hCG values that are within the range for pregnancy but are not pregnant (false positives) may be enrolled with written consent of the investigator, after pregnancy has been ruled out. Females of non-childbearing potential (postmenopausal for more than 1 year; bilateral tubal ligation; bilateral oophorectomy; hysterectomy) do not require a serum β-hCG test.
21. Women who are breastfeeding.
22. Patients who have prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's opinion, could affect the safety of the patient; alter the absorption, distribution, metabolism, or excretion of the study drug; or impair the assessment of study results.
23. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving Overall Response | Up to 12 months
  The overall response rate (ORR) will be defined as the number of evaluable patients whose best overall response to study treatment is complete response (CR) or partial response (PR). ORR will be assessed using Choi criteria by treating physician.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 years
  Progression-free survival (PFS) will be defined as the time elapsed from the start of treatment to the date of documented progression or death, whichever comes first. For surviving patients without progression who begin alternative treatment, PFS will be censored at the last date of documented progression-free status prior to starting alternative treatment. Similarly, losses to follow up will be censored at the last date of documented progression-free status.
Overall Survival (OS) | Up to 3 years
  Overall survival (OS) will be defined as the time elapsed from the start of treatment until death. For surviving patients, follow-up will be censored at the date of last contact.
Number of Participants Achieving Clinical Benefit | Up to 12 months
  The clinical benefit rate (CBR) will be defined as the number of evaluable patients whose best overall response to study treatment is complete response (CR), or partial response (PR), or stable disease (SD), for 6 months or more and will be assessed using Choi criteria by treating physician.
Incidence of Treatment-Related Toxicity and Adverse Events | Up to 13 months
  Safety and tolerability of assigned Sunitinib and Regorafenib treatment will be reported as the incidence of treatment-related toxicity, including serious adverse events (SAEs) and adverse events (AEs), in study participants using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Trent, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No